CLINICAL TRIAL: NCT00033696
Title: Paclitaxel/Topotecan/Etoposide (EtopoTax) Induction Followed by Consolidation Chemoradiotherapy for Limited Stage Small Cell Lung Cancer: A Phase II Study
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30002; U10CA031946 (NIH); CLB-30002; CDR0000069313 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; Carboplatin; Etoposide; Paclitaxel; Topotecan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy + radiation therapy (Experimental): Induction therapy: Patients receive paclitaxel IV over 3 hours on days 1 and 22, oral topotecan on days 2-4 and 23-25, and oral etoposide on days 5-7 and 26-28. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on days 8 and 29 and continuing until blood counts recover.
  Consolidation therapy: Patients receive carboplatin IV over 1 hour on days 43, 64, and 85 and etoposide IV over 1 hour on days 43-45, 64-66, and 85-87. Patients undergo radiotherapy daily 5 days per week beginning on day 43 and continuing for 6-7 weeks.
  Patients with rapid disease progression discontinue study therapy.
  Patients are followed at least every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: etoposide; Drug: paclitaxel; Drug: topotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: etoposide
Drug: paclitaxel
Drug: topotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and radiation therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete and overall response rates in patients with limited stage small cell lung cancer treated with induction chemotherapy comprising paclitaxel, topotecan, and etoposide followed by consolidation chemoradiotherapy.
* Determine the toxicity of this regimen in these patients.
* Determine the overall and failure-free survival of patients treated with this regimen.
* Determine the overall (partial and complete) response rate in patients treated with this induction chemotherapy regimen.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive paclitaxel IV over 3 hours on days 1 and 22, oral topotecan on days 2-4 and 23-25, and oral etoposide on days 5-7 and 26-28. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on days 8 and 29 and continuing until blood counts recover.
* Consolidation therapy: Patients receive carboplatin IV over 1 hour on days 43, 64, and 85 and etoposide IV over 1 hour on days 43-45, 64-66, and 85-87. Patients undergo radiotherapy daily 5 days per week beginning on day 43 and continuing for 6-7 weeks.

Patients with rapid disease progression discontinue study therapy.

Patients are followed at least every 3 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 25-60 patients will be accrued for this study within 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Limited stage defined as disease restricted to one hemithorax with regional lymph node metastases including hilar, ipsilateral, and contralateral mediastinal lymph nodes
* Measurable disease

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Lesions not considered measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions in a previously irradiated area
* No clinically suspected or confirmed supraclavicular lymph node metastases
* No pleural effusions visible on plain chest radiographs, regardless of cytology

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,00/mm3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT less than 2 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than ULN
* Creatinine clearance no greater than 150 mL/min for men or 130 mL/min for women

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other currently active malignancy except non-melanoma skin cancer
* Patients must have completed therapy for any other malignancy and be considered to be at less than 30% risk of relapse

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF) during consolidation therapy

Chemotherapy:

* No prior chemotherapy for small cell lung cancer
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except:

  * Steroids for adrenal failure
  * Hormones for non-disease-related conditions (e.g., insulin for diabetes)
  * Intermittent use of dexamethasone as an antiemetic or as an adjunct to prophylactic cranial irradiation

Radiotherapy:

* See Disease Characteristics
* No prior chest radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2001-09; Primary Completion 2007-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
overall response rate | up to 5 years

SECONDARY OUTCOMES:
failure-free survival | up to 5 years
overall survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonius A. Miller, MD, Study Chair — Wake Forest University Health Sciences
Locations (51):
- United States (51):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Miller AA, Wang XF, Bogart JA, Hodgson LD, Rocha Lima CM, Radford JE, Vokes EE, Green MR; Cancer and Leukemia Group B (CALGB). Phase II trial of paclitaxel-topotecan-etoposide followed by consolidation chemoradiotherapy for limited-stage small cell lung cancer: CALGB 30002. J Thorac Oncol. 2007 Jul;2(7):645-51. doi: 10.1097/JTO.0b013e318074bbf5. PMID 17607121